CLINICAL TRIAL: NCT00419653
Title: Modulation of Regional Brain Activation in Schizophrenic Patients by Pharmacological Therapy With Amisulpride, Olanzapine or Haloperidol. A Study With Functional Magnetic Resonance Imaging (fMRI) and Diffusion Tensor Imaging (DTI)
Brief Title: Modulation of Regional Brain Activation in Schizophrenic Patients by Pharmacological Therapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: University of Jena (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Dr. Ralf Schlösser, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia fMRI drug therapy amisulpride
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride; Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Amisulpride
- 2 (Active Comparator)
  Interventions: Drug: Olanzapine
- 3 (Active Comparator): Haloperidol
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Amisulpride
  Arms: 1
Drug: Olanzapine
  Arms: 2
Drug: Haloperidol
  Arms: 3

SUMMARY:
The study aims to investigate the modulation of regional brain activation in schizophrenic patients by psychopharmacological treatment with either haloperidol, amisulpride or olanzapine. The study will be performed with functional magnetic resonance imaging (fMRI) and diffusion tensor imaging (DTI).

DETAILED DESCRIPTION:
The current study aims to investigate the following issues:

* Changes in cognitive activation patterns under therapy with the typical neuroleptic haloperidol as compared to the atypical antipsychotics amisulpride and olanzapine
* Relationship of these changes in activity to psychopathological, neuropsychological and pharmacotherapeutic variables (e.g. drug plasma level) as well as to certain biological markers (HVA, prolactin)
* Relationship between diffusion anisotropy as an indicator for structural connectivity and cognitive activation patterns under antipsychotic treatment

ELIGIBILITY:
Inclusion Criteria:

* In- and outpatients of either sex
* Able to comply with the protocol
* Having given their written informed consent of their own free will
* Total BPRS (PANSS-derived, 1-7 points) minimum 36 points at baseline
* Schizophrenic or schizophreniform disorder according to DSM-IV criteria (295.10, .30, .40, .90)
* Definite right-handedness (according to the modified Edinburgh Handedness Inventory)
* Age 18 - 50 years

Exclusion Criteria:

* Co-morbid psychiatric axis I disorder (DSM-IV) other than schizophrenia
* Axis II disorder according to DSM-IV
* Present or past history of substance and drug dependence (including alcohol dependence)
* Participation in a clinical trial within the previous three months
* Lack of insight
* Suicidal ideations or aggression against others
* Consumption of caffeine-containing beverages within 6 hours before assessments
* Clinically significant findings in ECG or EEG
* Known intolerance against neuroleptics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Activation/deactivation in fMRI | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Schlösser, M.D., Principal Investigator — FSU Jena

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149